CLINICAL TRIAL: NCT05845502
Title: Single-arm, Open-label Clinical Study of SZ003 in the Treatment of Advanced Hepatocellular Carcinoma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Failed to recruit more volunteers
Sponsor: Shantou University Medical College (Other)
Collaborators: Guangdong ProCapZoom Biosciences Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yao KaiTao, Deputy Director, Shantou University Medical College
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PCZCTP-220808-001
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Advanced Hepatocellular Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SZ003 CAR-NK (Experimental)
  Interventions: Biological: SZ003 CAR-NK

INTERVENTIONS:
Biological: SZ003 CAR-NK — Drug: SZ003 CAR-NK In the escalation study, the minimum initial dose was 5.0×10^6 cells, then increased to 1.0×10^8 ,2.0×10^8 and5.0×10^8 cells. The infusion is given every 2 weeks.

SUMMARY:
This study was a single-center, open-label, investigator-initiated clinical trial (IIT) to observe and investigate the clinical safety and efficacy of SZ003 in the treatment of advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. With advanced hepatocellular carcinoma (HCC) confirmed by histopathology;
2. With stage C according to the Barcelona liver cancer grading criteria (BCLC) or with stage B who are ineligible for locoregional/locoregional therapy progression;
3. Unsuitable for surgery or local therapy (including ablation, interventional and radiotherapy) and who have experienced progression or intolerance after previous standard therapy;
4. Through immune tissues chemistry, confirmation of tumor cells positive expression of relevant molecular targets (GPC3) ;
5. With at least one stable evaluable target lesion according to RECIST 1.1 criteria, which was defined as: non-nodal lesion longest diameter ≥10 mm, or nodal lesion short diameter ≥15 mm;
6. Age 18-80, male or female;
7. Karnofsky Performance Status (KPS)≥80;
8. Stable vital signs and expected survival at least 12 weeks.
9. If HBsAg or HBcAb is positive, HBV-DNA < 200 IU/ml and to receive anti-HBV therapy ((Entecavir or tenofovirdisoproxil) for at least 14 days prior to the start of study treatment;
10. Blood Routine: WBC≥2.5×109/L, PLT≥60×109/L, Hb≥9.0g/dL, LY≥0.4×109/L;
11. Blood biochemistry: Alb≥30g/L, Lipase and Amylase ≤1.5 ULN, Serum creatinine ≤1.5 ULN, creatinine clearance ≥40mL/min, ALT≤5 ULN, AST≤5 ULN, Total Serum bilirubin ≤2.5 ULN, prothrombin time ≤6s;
12. Be able to understand and sign an informed consent form

Exclusion Criteria:

1. With uncontrolled active infections;
2. No other prior malignancy except nonmelanoma skin cancer or carcinoma in situ of the cervix within 5 years before study treatment initiation.
3. With previous history of encephalopathy.
4. With active acute or chronic virus, germ infection;
5. Diagnosed with HIV infection or active hepatitis, HBV, HCV infection or other serious infectious diseases;
6. Other serious medical conditions that may limit participation in the trial (such as poorly controlled diabetes (treated Glycated hemoglobin HbA1c > 7%) , severe heart failure (left ventricular ejection fraction (LVEF) < 45%) , myocardial infarction or unstable arrhythmia or unstable angina in the last 6 months, pulmonary embolism, chronic obstructive pulmonary disease, Interstitial lung disease, pulmonary function test FEV1 < 60% predicted, gastric ulcer, history of gastrointestinal bleeding, or definite gastrointestinal bleeding tendency) ;
7. Ascites more than 5cm;
8. The proportion of liver replaced by tumor≥70%, or with tumor infiltration in the portal vein, hepatic veins or inferior vena cava that completely blocks circulation in liver;
9. Prior solid organ transplantation or waiting for organ transplantation (including liver transplantation);
10. Prior anti-tumor therapies within 14 days before study treatment initiation, such as surgery, interventional therapy, radiotherapy, chemotherapy, immunotherapy.
11. Long-term systemic steroid therapy or patients with autoimmune diseases;
12. With a history of allergic reactions attributed to compounds of similar chemical or biological composition used in the study;
13. Have participation in clinical trials of any other investigational agents within 3 months before study treatment initiation.
14. Had received cell therapy previously but ineffective,after physical examination not allowed to received CAR-NK therapy by investigator's judgement;
15. Pregnant or lactating women;
16. Inappropriate to participate in this clinical trial by investigator's judgement.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2021-07-26 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
The incidence rates and severity of AEs | through study completion, an average of 1 year
  To evaluate the safety of SZ003 CAR-NK Cells

SECONDARY OUTCOMES:
overall survival (OS) | up to 2 years
  To determine the anti-tumor effectivity of SZ003 CAR-NK Cells
progression-free survival (PFS) | up to 2 years
  To determine the anti-tumor effectivity of SZ003 CAR-NK Cells
disease control rate (DCR) and objective response rate (ORR) | up to 2 years
  To determine the anti-tumor effectivity of SZ003 CAR-NK Cells
duration of response (DOR) | up to 2 years
  To determine the anti-tumor effectivity of SZ003 CAR-NK Cells

CONTACTS AND LOCATIONS:
Locations (1):
- Shantou University Medical College, Shantou, Guangdong, China